CLINICAL TRIAL: NCT04451902
Title: COVID-19 and Rare Skin Diseases. European Observational Study (Data Research) During an Epidemic
Brief Title: COVID-19 and Rare Skin Diseases European Observational Study During an Epidemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imagine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: COVID19-RareSkin
Record Dates: First submitted 2020-06-23; First posted 2020-06-30 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Rare Diseases
Keywords: skin
MeSH Terms: conditions — Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a European observational cohort study (data research) involving multiple centres to look at the potential impact of COVID infection on patients with rare skin diseases examining factors such as comorbidity, protection factors, and clinical and/or therapeutic factors. The data collected may provide additional information on the situation of patients and, on a wider basis, provide useful data applicable to the general population.

DETAILED DESCRIPTION:
Medical and demographic data will be collected from the medical records of patients. The data required will be specified in Appendix 1 (collection form). Patients will be identified by their initials (first letter of their surname and first name); The study will last for one year to cover the COVID-19 epidemic in France (which includes the areas of mainland France and its overseas departments and territories) and in Europe, via the ERN-Skin European Network.

The frequency of severe forms of COVID-19 will be calculated with a bilateral 95% confidence interval using, as a numerator, the number of patients with a severe form of COVID-19 and, as a denominator, the number of patients with a COVID-19 diagnosis confirmed by PCR, chest scan, serological assay or by suggestive clinical signs during the medical consultation. A severe form of COVID is defined as a case requiring hospitalisation in an intensive care unit, requiring resuscitation, or resulting in death.

Analysis of the impact of COVID-19 infection on rare skin diseases: complications, potential comorbidity factors, impact on the management of chronic conditions (change in treatment) and the experience of patients.

The results of the analysis may be compared with those obtained for other groups of diseases. Gaining a better understanding of high-risk situations, as well as any aggravation or protective factors, should enable us to issue recommendations adapted to this kind of disease but that may also be useful for the general population. This type of study may also provide "reassurance" to patients with rare diseases who have many questions during this period of epidemic and heightened concern.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a rare skin disease,
* Patient of any age (paediatric or adult),
* Patient with suspected COVID-19 infection (remote consultation, face-to-face consultation, general practitioner, hospital physician),
* Patient in contact with a subject infected with the COVID-19 virus,
* Asymptomatic patient for COVID-19 viral infection but with a positive serology,
* Study information given to the patient and/or to their legal representative,
* Patient who has been informed and has agreed to this data collection process.

Exclusion Criteria:

* Patients not suffering from a rare skin disease,
* Patient and/or their legal representative who object to their participation in the study at the presentation of the information leaflet,
* Adult patient unable to understand the implications and constraints of the study,
* Protected adult subject to guardianship or safeguarding measures.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a European observational cohort study (research data) involving multiple centres whose main objective is to determine the impact of a COVID-19 virus infection in a cohort of patients with rare skin diseases and particularly if these rare diseases and their treatments are risk factors of infection severity. The cohort of patients with rare skin diseases is monitored by the European Reference Network (ERN-Skin) and FIMARAD network centres. This is a public health impact study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Analysis of the impact of COVID-19 infection on rare skin diseases: complications | Baseline
  Frequency of hospitalisations related to suspected and confirmed cases of Covid-19 infection and consequences
Analysis of the impact of COVID-19 infection on rare skin diseases: potential comorbidity factors | Baseline
  Frequency of hospitalisations related to suspected and confirmed cases of Covid-19 infection and analysis of associated factors: age, gender, pathology, comorbidities, medications
Analysis of the impact of COVID-19 infection on rare skin diseases: impact on the management of chronic conditions (change in treatment) | Baseline
  Frequency of confirmed and suspected unconfirmed Covid-19 infections; description of clinical signs and signs of an impact on the chronic disease; description of possible therapeutic changes due to the Covid-19 infections

CONTACTS AND LOCATIONS:
Overall Officials: Christine BODEMER, Principal Investigator — Hôpital Necker-Enfants Malades
Locations (13):
- University Hospital Brno - EB Centrum CR Dermatolog, Brno, Czechia
- France (6):
  - Hôpital de l'Archet 2 (CHU de Nice), Nice, Alpes-Maritimes
  - Hôpital de Clocheville (CHRU de Tours), Tours, Indre-et-Loire
  - Hôpital de Brabois (CHU de Nancy), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hôpital Charles Nicolle (CHU de Rouen), Rouen, Seine-Maritime
  - Hôpital Saint Louis (AP-HP), Paris, Île-de-France Region
  - Hôpital Necker - Enfants malades (AP-HP), Paris, Île-de-France Region
- Germany (2):
  - University Hospital of Erlangen - ZSEER - Zentrum für Seltene Erkrankungen Erlangen, Erlangen, Bavaria
  - Städtisches Klinikum Dessau, Dessau Medical Center, Dessau, Saxony-Anhalt
- Italy (3):
  - Istituto Dermopatico dell'Immacolata, Rome, Lazio
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda USL Toscana Centro, Florence, Tuscany
- Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas, Lithuania